CLINICAL TRIAL: NCT07051876
Title: The Effects of Mouthguard and Physiotherapy on Bruxism: An EMG and Posture Angle Analysis
Brief Title: Feasibility of a Clinical Trial on Physiotherapy and Mouthguards for Bruxism Using Posture and EMG Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Usj-2023-200
Record Dates: First submitted 2025-04-16; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Bruxism; Manual Theapy
MeSH Terms: conditions — Bruxism | interventions — Mouth Protectors; Physical Therapy Modalities; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mouthguard Only (Experimental): participants in this arm receive a custom-fitted thermoplastic mouthguard (3A MEDES®) fabricated by a dentist. The mouthguard is worn nightly during sleep for 6 weeks. Participants are instructed on daily cleaning and proper storage. No additional treatments are provided in this arm.
  Interventions: Device: Mouthguard Only
- Mouthguard and Physiotherapy (Experimental): Participants in this arm receive the same custom-fitted mouthguard as in the first arm, worn nightly for 6 weeks, along with a daily home-based physiotherapy protocol that includes:
  Postural correction exercises
  Mandibular awareness training
  Relaxation techniques (e.g., Bae method)
  Diaphragmatic breathing (5 minutes daily or 15 repetitions)
  Self-massage of masseter and temporalis muscles
  Stretching and jaw coordination exercises
  Jaw muscle strengthening with resistance
  Participants perform exercises once daily for 6 weeks and submit daily video recordings via a messaging platform (e.g., Teams or WhatsApp) to ensure compliance.
  Interventions: Device: Mouthguard and Physiotherapy

INTERVENTIONS:
Device: Mouthguard and Physiotherapy — The mouthguard and physiotherapy group will receive a custom-fitted mouthguard along with a physiotherapy program. The home-based physiotherapy exercises will include posture improvement routines, relaxation techniques, and targeted therapy for the muscles of the head, neck, and shoulders. These sessions will be performed daily at home for a duration of six weeks. Each participant will sign a consent form approved by the Ethics Committee of Saint Joseph University.
  Other Names: MANUAL THERAPY; MOUTHGUARD
  Arms: Mouthguard and Physiotherapy
Device: Mouthguard Only — The mouthguard only group will receive a custom-fitted mouthguard, which will be fabricated by a qualified dentist. The mouthguard will be worn during sleep for 6 weeks. Participants will be instructed to clean the mouthguard daily and to store it in a cool, dry place.
  Arms: Mouthguard Only

SUMMARY:
The purpose of this research is to determine whether a clinical trial assessing the impact of physiotherapy and mouthguards on bruxism is feasible. This includes evaluating the feasibility of participant recruitment, implementing the interventions, and collecting data using appropriate techniques. The study will focus on posture angle analysis to assess changes in posture associated with bruxism, and electromyography (EMG) to measure muscular activity. By examining these elements, the study aims to lay the groundwork for a larger clinical trial that could provide conclusive evidence regarding the efficacy of these therapies in treating bruxism.

Participants will be recruited from the USJ dental clinics following their consultation. They will be screened for bruxism using a questionnaire and a clinical examination based on the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).

The mouthguard-only group will receive a custom-fitted mouthguard, fabricated by a qualified dentist. Participants will be instructed to wear the mouthguard during sleep for six weeks, to clean it daily, and to store it in a cool, dry place.

The mouthguard and physiotherapy group will receive both a custom-fitted mouthguard and physiotherapy. The home physiotherapy program will include posture improvement exercises, relaxation techniques, and muscle therapy targeting the head, neck, and shoulders. Participants will perform the exercises daily at home, record themselves, and submit the videos each day via a social platform (e.g., Microsoft Teams or WhatsApp, depending on patient preference) for a period of six weeks.

DETAILED DESCRIPTION:
Participant recruitment was conducted at USJ dental clinics with support from the occlusal department and private clinic following patient consultations. Screening for bruxism involved a clinical examination and the DC/TMD questionnaire. Ethical approval was granted by the Saint Joseph University of Beirut (approval number USJ-2023-200), and informed consent was obtained from all participants.

Electromyographic (EMG) assessments were carried out by the principal investigator using a portable EMG machine (KM560). Electrodes were placed bilaterally on the masseter muscles. Participants were instructed to bite in maximum intercuspation six times for five seconds each, with rest intervals in between. The device recorded muscle activity during both contraction and relaxation phases to evaluate bruxism-related muscle function.

Forward head posture was analyzed through photogrammetry. Markers were placed at the tragus of the ear and the C7 vertebra. Lateral photographs were taken, and the craniovertebral angle was measured using image analysis software to assess postural alignment.

The physiotherapy protocol consisted of a six-week home program performed daily. It included awareness of the mandibular rest position, relaxation techniques, diaphragmatic breathing, self-massage of the masseter and temporalis muscles, stretching, coordination, and resistance exercises. Participants recorded and submitted daily videos via Teams or WhatsApp to ensure compliance.

Custom mouthguards were fabricated by the researcher. Dental impressions were taken using alginate (Hydrogum 5®), and casts were made. Mouthguards were then vacuum-formed using thermoplastic material (3A MEDES®), followed by trimming and polishing to ensure a comfortable fit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Confirmed diagnosis of bruxism by a qualified member of the occlusion unit department
* No history of temporomandibular disorders or other craniofacial pain conditions
* No history of neurological or psychiatric disorders
* No current use of medications that affect muscle tone or sleep

Exclusion Criteria:

* - The presence of any systemic or neuromuscular disorder affecting the jaw muscles or posture.
* Use of medications, substances, or drugs that may affect jaw muscle activity, such as muscle relaxants or stimulants.
* Lifestyle: sleep disorder, anxiety
* Presence of any oral pathology or dental prostheses that may interfere with the use of a mouthguard.
* Inability to tolerate the EMG electrodes or posture angle analysis.
* Patient who has recently undergone physiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Change in Masseter Muscle Activity and Cervical Posture Angle from Baseline to 6 Weeks Measured by Surface EMG and Postural Assessment Tools. | From enrollment to the end of treatment at 6weeks
  Surface electromyography (sEMG) will be used to measure muscle activity of the masseter and temporalis during rest and clenching. A posture assessment tool will evaluate changes in head and cervical posture using digital angle measurements. Measurements will be taken at baseline and after 6 weeks of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph university, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barros Vde M, Seraidarian PI, Cortes MI, de Paula LV. The impact of orofacial pain on the quality of life of patients with temporomandibular disorder. J Orofac Pain. 2009 Winter;23(1):28-37. PMID 19264033